CLINICAL TRIAL: NCT05597969
Title: The Effect of an Application-based Health Intervention (FoodCoach) on Food Purchases in Switzerland: Randomized Controlled Trial
Brief Title: The Effect of an Application-based Health Intervention (FoodCoach) on Food Purchases in Switzerland
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of St.Gallen (Other)
Collaborators: University hospital of Bern (Unknown); Swiss National Science Foundation (Other); Sanitas Management AG (Unknown)
Responsible Party: Principal Investigator, Wu Jing, PhD Candidate and Project Leader, University of St.Gallen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FOODCOACH2022
Record Dates: First submitted 2022-10-21; First posted 2022-10-28 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Adult
Keywords: eHealth; Food purchase; Behavior change; Randomized controlled trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FoodCoach (Experimental): The experimental group uses the FutureMe app for 9 weeks and continue to voluntarily use it. The app has the following functionality:
  * Dashboard: show the Nutri-Score changes over the last 10 baskets and comparisons between the specific user and all FoodCoach app users.
  * Recommendations: show three recommendations regarding their food purchases and healthier product recommendations to help them achieve these recommendations.
  * Nutrition Analysis: show the monthly energy contribution of 7 food categories in the past 6 months.
  * Spending Analysis: show the monthly expense contribution of 7 food categories and 1 not categorized category in the past 6 months.
  * Shopping history: show their purchase history in the past 6 months, together with monthly average Nutri-Score and basket Nutri-Score if applicable
  * Q & A: show answers to the commonly asked questions. E.g., how is the Nutri-Score calculated?
  Interventions: Behavioral: FoodCoach
- Control (No Intervention): The control group receives no application for use. They need to finish the onboarding survey, donate their food purchase data and finish the post-study survey (voluntary). They receive no intervention while the experimental group should be actively using the FoodCoach app. The investigators will send them an analysis report of their food purchase data via email in 3 months after the intervention phase is gone. Note the intervention lasts for 9 weeks.

INTERVENTIONS:
Behavioral: FoodCoach — The FoodCoach app displays transparent analysis and recommendations regarding participant's food purchases recorded on their loyalty cards. It tries to help participants understand why and how they should/can shop more healthily, motivating them to change their unhealthy food purchase behavior.
  Arms: FoodCoach

SUMMARY:
The FoodCoach study is a 9-week randomized controlled trial from the University of St.Gallen and the University Hospital of Bern, supported by the Swiss National Science Foundation #188402 and by Sanitas Management AG. Sanitas Management AG supports the recruiting of study participants without interfering with the study content.

FoodCoach aims to investigate the effectiveness of improving people's food shopping healthiness by providing automated food shopping recommendations. The results of the study could possibly help improve the health status of the Swiss population and beyond in a low-cost and automated manner.

The investigators collect participant grocery data via the loyalty card programs "Migros Cumulus" and "Coop Supercard" after obtaining participants' informed consent. From this data, the investigators generate automated recommendations that are based on the Nutri-Score framework and expertise of dieticians at the University Hospital of Bern. After sign-up, participants are randomized into a treatment and a control group. The treatment group receives automated recommendations via the FoodCoach Web Application, while the control group only receives a report about their food shopping by email after the intervention phase. Both groups need to finish the same onboarding survey where the investigators collect basic demographic information. After the intervention, the treatment group will receive a post-study survey containing two parts via email. Part 1 includes questions about the ease of use, interface and satisfaction and usefulness of the FoodCoach app. Part 2 includes questions about the participants' weight and height, the motivation to shop healthily and sustainably. The control group will receive a post-study survey which only contains part 2 as described before via email.

ELIGIBILITY:
Inclusion Criteria:

* Participants need to be at least 18 years old by the time they join the study.
* Participants need to participate in at least one of the two loyalty card programmes, i.e., Migros Cumulus and/or Coop Supercard.
* Participants need to be German- and/or English-speaking, as the FoodCoach application is in German and English.

Exclusion Criteria:

* Younger than 18 years old by the time the participants join the study.
* Do not participate in at least one of the two loyalty card programmes, i.e., Migros Cumulus and/or Coop Supercard.
* Not German- and/or English-speaking, so that the participants cannot understand the content of the app.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Body mass index change | Baseline, 9 weeks
  Survey data. Note that the post-study survey is "voluntary" because the investigators cannot force participants to finish it.
Food purchase behavior - overall food shopping healthiness change | Baseline, 9 weeks
  The overall food shopping healthiness as indicated by Food Standards Agency Nutrient Profiling System Dietary Index
Food purchase behavior - fruit purchase change | Baseline, 9 weeks
  Loyalty card data
Food purchase behavior - vegetable purchase change | Baseline, 9 weeks
  Loyalty card data
Food purchase behavior - protein food purchase change | Baseline, 9 weeks
  Loyalty card data
Food purchase behavior - processed food purchase change | Baseline, 9 weeks
  Loyalty card data
Food purchase behavior - beverage purchase change | Baseline, 9 weeks
  Loyalty card data
Food purchase behavior - oils, fats, sauces, nuts and seeds purchase change | Baseline, 9 weeks
  Loyalty card data
Food purchase behavior - grains, potatoes and legumes purchase change | Baseline, 9 weeks
  Loyalty card data

SECONDARY OUTCOMES:
Food purchase behavior - energy purchase change | Baseline, 9weeks
  Loyalty card data
Food purchase behavior - sugar purchase change | Baseline, 9weeks
  Loyalty card data
Food purchase behavior - saturated fatty acids purchase change | Baseline, 9weeks
  Loyalty card data
Food purchase behavior - sodium purchase change | Baseline, 9weeks
  Loyalty card data
Food purchase behavior - fiber purchase change | Baseline, 9weeks
  Loyalty card data
Food purchase behavior - protein purchase change | Baseline, 9weeks
  Loyalty card data

CONTACTS AND LOCATIONS:
Overall Officials: Jing Wu, MSc., Principal Investigator — University of St.Gallen
Locations (1):
- University of St. Gallen, Sankt Gallen, Canton of St. Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
We plan to published anonymized partial food purchase data as approved by the Ethics committee.
  1. The data will be published in an anonymized form.
  2. Only purchase records that can be identified by our food composition database and belong to certain food categories will be published.
Supporting Information: SAP, ICF
Time Frame: The data will become available in 2023, published together with the corresponding paper to ensure the results are reproducible. It will be available until participants request to delete their data.